CLINICAL TRIAL: NCT01778699
Title: Anticaries Effect of Probiotic Lactobacillus Brevis CD2 (Lb CD2). A Randomized Double Blind Interventional Study.
Brief Title: Anticaries Effect of Probiotic Lactobacillus Brevis CD2 (Lb CD2).
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: University of Milan (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Guglielmo Campus, Associate Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013_01_21_a
Record Dates: First submitted 2013-01-21; First posted 2013-01-29 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Dental Caries; Gingivitis
Keywords: Lactobacillus brevis CD2; caries incidence; plaque-pH
MeSH Terms: conditions — Dental Caries; Gingivitis | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lozenges with Lactobacillus brevis CD2 (Experimental): During the treatment phases subjects will use 2 lozenges a day.
  Interventions: Dietary Supplement: lozenges
- Lozenges (Placebo Comparator): During the treatment phases subjects will use 2 lozenges a day.
  Interventions: Dietary Supplement: lozenges

INTERVENTIONS:
Dietary Supplement: lozenges — The test products for the study is manufactured and provided by CD Investments srl, Italy. The placebo lozenges will look like the active lozenges with the same taste and weight of 1 gram containing only the ingredients listed above in the same proportion as the active but with no L. brevis CD2. It will not be possible to differentiate the two products.
  The study center and the monitor must be informed of any deficiency in the study products (products will be kept at 4° degrees during the study).

SUMMARY:
In a previous study the efficacy of Lb CD2 on interim covariates related to caries development was tested. So, it was decided to plan a new study on schoolchildren from the same area. The aim of the present research protocol was to evaluate the anticariogenic effect of probiotics daily used, on the caries development in children. The null hypothesis was that the probiotic Lb CD2 would not modify the caries risk of the children. Moreover, the study will be carried out to investigate the plaque acidogenicity in situ following the regular consumption of a probiotic product compared to a control group.

Objective: To determine the effect of a regularly consumed probiotic on the development of new caries lesions.

Study design: Double blind, placebo-controlled, longitudinal study, monocentric, national, in situ

DETAILED DESCRIPTION:
2 RATIONALE FOR THE STUDY In a previous study the efficacy of Lb CD2 on interim covariates related to caries development was tested. So, it was decided to plan a new study on schoolchildren from the same area. The aim of the present research protocol was to evaluate the anticariogenic effect of probiotics daily used, on the caries development in children. The null hypothesis was that the probiotic Lb CD2 would not modify the caries risk of the children. Moreover, the study will be carried out to investigate the plaque acidogenicity in situ following the regular consumption of a probiotic product compared to a control group.

3 STUDY OBJECTIVES

Primary objective:

The regular consumption of probiotic will lead to a significantly lower caries increment compared to a placebo. Regular oral hygiene is permitted.

.

Target criteria:

Efficacy: Lower caries increment Safety: Determination of side effects

Safety: Determination of side effects Side effects such an especially changes of the oral mucosa after the consumption of the product.

4 STUDY DESIGN 4.1 Study design and study centre Double blind, placebo-controlled, longitudinal study on 440 test subjects. The study will be carried out at a single centre in the Department of Surgery, Microsurgery and Medical Sciences -School of Dentistry of the University of Sassari, Viale San Pietro 43/C Sassari.

The planned duration of the study is January-February 2013 to March 2015 (with Final Report).

Proposed start of the recruitment of test subjects January-February 2013.

5 TEST SUBJECTS 440 healthy male or female chidren test subjects. These will be recruited from primary schools in Sassari.

5.1 Concomitant treatment not permitted In general, other probiotic-containing products, except dairy products.

5.2 Permitted concomitant medication All other medications are allowed. However, for the 30 days prior to the screening phase and during the entire study period, they must be entered in the case report form under the "Concomitant Medication" section.

5.3 Criteria for premature termination of the study in individual test subjects.

Reasons which may be given for the premature withdrawal of an individual test subject are:

* Retraction of consent
* If continued participation in the study is no longer acceptable or justified on important medical grounds as assessed by the investigator
* Occurrence of intolerable side effects (SE) as assessed by the investigator
* Violation of the protocol, according to the decision of the investigator, with reasons given in writing
* Non-attendance by the test subject
* Lack of compliance and motivation on the part of the test subject (e.g. not wearing the intra-oral specimen holder for more than six hours a day) Test subjects who withdraw from the study prematurely should be subjected to the final examination.

The reasons for withdrawal from the study and the date must be recorded by the investigator in the case report form.

5.4 Criteria for discontinuing the entire study In particular, the recognition of new information and/or risks which requires the benefit/risk ratio to be reassessed. In the case of a negative outcome, the LKP may discontinue the study in discussion with the principal investigator and the sponsor.

If there is inadequate recruitment or persistent or recurrent serious objection to the trial protocol, the sponsor, in agreement with the LKP and after discussion with the principal investigator, may decide to terminate the study prematurely for administrative reasons.

Should the premature termination of the study be unavoidable, measures must be decided upon and introduced to protect the interests and well-being of the test subjects as far as possible.

6 STUDY PRODUCTS 6.1 Test products and placebo The test products for the study is manufactured and provided by CD Investments srl, Italy. The placebo lozenges will look like the active lozenges with the same taste and weight of 1 gram containing only the ingredients listed above in the same proportion as the active but with no L. brevis CD2. It will not be possible to differentiate the two products.

The study center and the monitor must be informed of any deficiency in the study products (products will be kept at 4° degrees during the study).

6.2 Standard toothpaste and toothbrushes Standard toothpaste containing fluoride: monofluorophosphate containing toothpaste (800/1000 ppm)

6.3 Packaging and labelling 6.3.1 Test product Before use, the investigator will store the test samples at 4° degrees temperature. For each subject one container of study medication for the study period will be delivered, as well as one replacement container in each case. The test samplesy were produced and supplied by CD investiments (Italy) and coded as either 'green' or 'red'. The code was sealed by an independent monitor, and not broken until the statistical analysis was finalized.

6.4 Determination of compliance 6.4.1 Test medication The containers will be weighed before and after the study period.

6.4.2 Standard toothpaste The test subjects must use the standard toothpaste throughout the study. A check will be made on compliance by questioning the test subject.

6.5 Documentation on the whereabouts of the test samples The investigator will record the whereabouts of the test samples in an inventory. Delivery notes and notices of returns will be signed by the investigator.

7 DOSAGE In the treatment phase subjects will use 2 losanges a day.

8 STUDY SCHEDULE AND TEST METHODS 8.1 Study schedule 8.1.1 Planned schedule Prior to the start of the study, demographic, ethnic and prognostic data will be collected (screening phase). A medical history will be taken, with documentation of previous and concomitant treatment and a clinical examination of the oral cavity (dental status, oral mucosa) will be performed by the investigator. If the test subject meets all the inclusion criteria without fulfilling any of the exclusion criteria, he/she will be enrolled in the clinical trial and given a test subject identification number.

All test subjects will receive a patient diary in the screening phase. Individual specimen holders will now be prepared for each test subject.

Period 1: (180 days) consumption of the study product, regular oral hygiene At the start of the period ICDAS score will be recorded with plaque pH and salivary mutans streptococci. All subjects are instructed about oral hygiene and about the consumption of the study product. At the 90th day plaque pH and salivary mutans streptococci will be also recorded again.

Period 2: (90 days) regular oral hygiene plaque pH and salivary mutans streptococci will be recorded again. Period 3: (180 days) consumption of the study product, regular oral hygiene At the start of the period ICDAS score will be recorded with plaque pH and salivary mutans streptococci. All subjects are instructed about oral hygiene and about the consumption of the study product. At the 90th day plaque pH and salivary mutans streptococci will be also recorded again.

Period 4: (90 days) regular oral hygiene plaque pH and salivary mutans streptococci will be recorded again. Period 5: (180 days) consumption of the study product, regular oral hygiene At the start of the period ICDAS score will be recorded with plaque pH and salivary mutans streptococci. All subjects are instructed about oral hygiene and about the consumption of the study product. At the 90th day plaque pH and salivary mutans streptococci will be also recorded again.

9 MATERIALS AND METHODS 9.1 Clinical parameters ICDAS (International Caries Detection and Assessment System) index, Oral mucosa

9.2 Investigation of saliva factors Saliva factors pH and flow rate will be measured during the screening phase on three days, each time in the morning. The mean of the three measurements will be calculated.

The Dentobuff® test kit (Vivadent, Liechtenstein) will be used.

9.3 Teeth brushing technique Test subjects are required to clean their teeth at minimum two times a day with the fluoride-containing toothpaste and a soft toothbrush. During that time, a fresh, damp gauze (soaked in water) will be placed in the container each day in order to provide a moist atmosphere for the appliances. The specimens should not be allowed to dry out.

The enamel specimens themselves are likewise carefully cleaned with the soft toothbrush except the last day of every period.

9.4 Randomization Using a computer program (Excel 2010 for Mac OsX), the randomization will carried out on an individual basis.

9.5 Application of the study product The subjects are not allowed to chew the lozenges. They are allowed to swallow the lozenges.

9.6 Plaque-pH evaluation At the end of each phase plaque acidogenicity will be assessed using the MicroTouch technique after a previous sucrose challenge. Evaluations of pH will be carried out at on each specimen. The pH will be measured in quintuplicate at 6 different time points: at baseline (before sucrose rinse) and 2, 5, 10, 20 and 30 min after a 1-min rinse with 10 ml 10% sucrose, using active movements.

An iridium touch microelectrode (diameter 0.1 mm; Beetrode NMPH-1, World Precision Instruments, Sarasota, Fla., USA, with a porous glass reference electrode (MERE 1, World Precision Instruments) will be used. A salt bridge will be created in a KCl (3 M) solution between the reference electrode and a finger of the subject. Before each session of pH evaluation, the electrode will be calibrated using buffer solution at pH 7.00 and 4.00.

ELIGIBILITY:
Inclusion Criteria:

* Written declaration of informed consent signed by parents/guardian
* At least 20 teeth
* Good general health, as assessed by investigator
* Average oral hygiene (cleaning the teeth at least twice a day)
* Agreement of test subject not to use any oral hygiene products other than the test products and toothpaste provided for the duration of the study; the use of non-fluoridated oral hygiene agents is allowed.
* Flow rate of stimulated saliva ≥ 0.7 ml/min
* High caries risk following Cariogram [Campus et al., 2009]

Exclusion Criteria:

* Ongoing oral or dental treatment except for emergency treatment.
* Known allergic reaction to an oral hygiene product and/or medication and/or dental material previously used in the mouth or pharynx.
* Existing allergy to one of the components of the test products or the standard toothpaste.
* Pathological changes of the oral mucosa, e.g. acute ulcerating gingivitis, acute herpetic gingivostomatitis, recurrent aphthous ulceration or systemic illnesses with oral manifestations.
* Antibiotic therapy within the past six months, used for a period more than 10 days.
* Any non-permitted therapy.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Caries increment by ICDAS method | 180 days
  ICDAS (International Caries Detection and Assessment System) index, Oral mucosa

SECONDARY OUTCOMES:
salivary mutans streptococci | 90 days
  Saliva factors and flow rate will be measured each time in the morning.
plaque pH | 90 days
  plaque pH after a rinse with a 10% sucrose solution for 1 min. Measurements of plaque pH will be performed before and after 2, 5, 10, 15 and 30 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Microsurgery and Medicine Sciences -School of Dentistry University of sassari, Sassari, SS, Italy